CLINICAL TRIAL: NCT07295626
Title: Effects of Reflexology Applied to Stroke Patients on Pain, Physiological Parameters and Sleep Quality: A Randomized Controlled Trial
Brief Title: Symptom Control and Physiological Effects of Reflexology Applied After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hakkari Universitesi (Other)
Responsible Party: Principal Investigator, Samet Koltaş, LECTURER, Hakkari Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HU-SHMYO-SK-01
Record Dates: First submitted 2025-11-23; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pain; Stroke; Reflexology; Nursing; Sleep Quality; Physiological Parameter
Keywords: pain; stroke; reflexology; nursing; sleep quality; Physiological Parameter
MeSH Terms: conditions — Pain; Stroke; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study was conducted using a randomized controlled intervention design. Participants were randomly assigned to the intervention and control groups. The intervention group received reflexology massage along with routine nursing care; the control group received only routine nursing care. During the intervention period, patients' pain levels, physiological parameters, and sleep quality were measured. Analyses were performed using appropriate statistical methods to evaluate differences between groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - Routine Care (No Intervention): This arm receives routine nursing care only, without reflexology massage. Physiological parameters, pain, and sleep quality are monitored twice weekly for six weeks, but no additional interventions are applied. This group serves as a comparison to evaluate the effects of reflexology.
- Reflexology Intervention Group (Experimental): This arm receives routine nursing care along with reflexology massage. Reflexology is applied twice a week for six weeks, with each session lasting 30 minutes (15 minutes per foot). The intervention aims to evaluate its effects on pain, physiological parameters, and sleep quality in stroke patients.
  Interventions: Other: Reflexology Intervention Group

INTERVENTIONS:
Other: Reflexology Intervention Group — This arm receives routine nursing care along with reflexology massage. Reflexology is applied twice a week for six weeks, with each session lasting 30 minutes (15 minutes per foot). The intervention aims to evaluate its effects on pain, physiological parameters, and sleep quality in stroke patients.
  Arms: Reflexology Intervention Group

SUMMARY:
This study is designed as a randomized controlled intervention with a pre-test-post-test design to evaluate the effect of reflexology on pain, physiological parameters, and sleep quality in stroke patients. The study will be conducted at the Physical Therapy and Rehabilitation Unit of Van Training and Research Hospital between October 2024 and June 2025.

Using a simple randomization method, patients will be assigned to either the control group or the reflexology intervention group, with an anticipated sample size of 35 patients per group. Data will be collected using the Personal Information Form, the Visual Analog Scale (VAS), the Richards-Campbell Sleep Scale (RCSS), and a physiological parameters recording form.

Patients in the intervention group will receive reflexology massage twice a week for six weeks, for a total of 12 sessions. Each session will last 30 minutes (15 minutes per foot), in addition to routine nursing care. Physiological parameters will be recorded before and after each reflexology session. The control group will receive routine nursing care only, and their physiological parameters will be monitored twice weekly using the same schedule. All scales and forms will be administered again at the end of the 6-week period.

The study aims to determine whether reflexology influences pain levels, physiological parameters, and sleep quality in stroke patients. Findings from this research may contribute to the evidence base regarding complementary interventions in post-stroke nursing care; however, no study results are yet available in this protocol record.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled experimental trial to evaluate the effects of reflexology applied to individuals who have experienced a stroke on pain levels, physiological parameters, and sleep quality. The study includes an intervention group and a control group and aims to examine the role of reflexology within a holistic nursing care approach.

The research will be conducted between October 2024 and June 2025 at the Physical Therapy and Rehabilitation Unit of Van Training and Research Hospital. A single-blind method will be used, in which information about group assignment will be concealed from participants. Ethical committee approval has been obtained from a foundation university, and institutional approval has been received from the hospital where the study will take place.

Using a simple randomization method, patients will be assigned to either the reflexology group or the control group, with an anticipated sample size of 35 participants in each group. Data will be collected using the Personal Information Form, the Visual Analog Scale (VAS), the Richards-Campbell Sleep Scale (RCSS), and a physiological parameters recording form.

Participants in the intervention group will receive reflexology massage twice a week for six weeks, for a total of 12 sessions, each lasting 30 minutes (15 minutes per foot), in addition to routine nursing care. Physiological parameters will be recorded before and after each reflexology session. Participants in the control group will receive routine nursing care only, and their physiological parameters will be monitored twice weekly following the same schedule. All forms and scales will be administered again at the end of the sixth week.

This study aims to determine whether reflexology has an effect on pain, physiological parameters, and sleep quality in individuals who have experienced a stroke. The findings of the study will contribute to the evidence base regarding complementary practices used in nursing care; however, no study results are reported in this protocol record.

ELIGIBILITY:
Inclusion Criteria:

Individuals over the age of 18,

* No diagnosis of any psychiatric illness or medication use,
* Hemiplegic stroke patients,
* Volunteering to participate in the study,
* According to the patient introduction form; patients describing hemiplegic shoulder pain and insomnia symptoms,
* No history of neurological or psychiatric disorders other than stroke,
* No irritation or ulceration in the skin area where reflexology will be performed,
* No history of deep vein thrombosis,
* Able to speak and understand Turkish and able to read and write,
* Patients who voluntarily agree to participate in the study will be included.

Exclusion Criteria:

Refusal to participate in the study,

* Tetraplegic and paraplegic patients,
* Patients with stroke due to malignant brain damage undergoing chemotherapy or radiotherapy
* Those with mental and psychiatric disorders,
* Those who have received professional massage therapy within the past month,
* Those with contraindications for foot massage and reflexology: patients with generalized edema, pacemakers, history of heart attack, active gout, history of deep vein thrombosis, history of gallbladder and kidney stones, acute infection, fever, fractures, or wounds will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline and at the end of week 6.
  Visual Analog Scale Pain intensity will be measured using the Visual Analog Scale, a 10-cm scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain, with higher scores reflecting greater pain intensity. VAS scores will also be classified as follows: 0 = no pain; 1-2 = very mild pain; 3-4 = mild pain; 5-6 = moderate pain; 7-8 = severe pain; 9-10 = very severe pain. This measure will be used to evaluate the effect of the reflexology intervention on pain levels in stroke patients, assessed at baseline and at the end of Week 6.

SECONDARY OUTCOMES:
Sleep Quality | Baseline and at the end of week 6.
  Richards Campbell Sleep Scale On the scale, where each sleep statement is scored from 0 to 100, "0" corresponds to the worst situation for each statement, and "100" corresponds to the best situation. As the score on the scale increases, sleep quality improves.
Systolic Blood Pressure | Before and after each reflexology session, twice weekly for 6 weeks.
  Systolic blood pressure will be measured in millimeters of mercury (mmHg) to evaluate changes associated with the reflexology intervention in stroke patients.
Diastolic Blood Pressure | Before and after each session, twice weekly for 6 weeks.
  Diastolic blood pressure will be measured in millimeters of mercury (mmHg) to assess physiological response to the reflexology intervention.
Heart Rate | Before and after each session, twice weekly for 6 weeks.
  Heart rate will be measured in beats per minute (bpm) to evaluate autonomic responses associated with the reflexology intervention.
Oxygen Saturation | Before and after each session, twice weekly for 6 weeks.
  Oxygen saturation will be measured using pulse oximetry and recorded as a percentage (%) to monitor potential changes associated with the reflexology intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Samet KOLTAŞ, Principal Investigator — Hakkari Universty
Locations (1):
- University of Health Sciences Van Training and Research Hospital, Van, Edremit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
individual participant data will be shared with other researchers. Data will be anonymized to protect participant privacy, and access will be provided upon request under specified conditions.
Time Frame: Individual participant data will be made available beginning 6 months after study completion and will remain accessible for a period of 5 years.
Access Criteria: Access to the de-identified individual participant data will be granted to qualified researchers who provide a methodologically sound research proposal and obtain ethics committee approval. Requests must include a brief study plan and justification for the use of the data. Data will be shared through secure institutional channels upon approval by the principal investigator and the hosting institution.

REFERENCES:
- See also: University of Health Sciences Van Training and Research Hospital — https://vaneah.saglik.gov.tr/TR
- See also: Hasan Kalyoncu University Faculty of Health Sciences — https://sbf.hku.edu.tr/

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-08-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT07295626/Prot_ICF_000.pdf